CLINICAL TRIAL: NCT00536978
Title: T-Cell or Natural Killer (NK) Cell Adback in Patients With Lymphoid Malignancies Receiving Allogeneic Stem Cell Transplantation With Campath-IH Containing Conditioning Regimens
Brief Title: Natural Killer (NK) Cell Adback After Allogeneic Stem Cell Transplant With Campath-IH Plus Chemorx for Patients With Lymphoid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0230
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Results first posted 2012-05-22 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Lymphoma; Leukemia
Keywords: Lymphoma; Leukemia; B-Cell Lymphoid Malignancies; CLL; Cll/Small Lymphocytic Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Diffuse Large Cell Lymphoma; Splenic Lymphoma; MALT; Lymphoplasmacytic Lymphoma; Burkitt's Lymphoma; ARA-C; BCNU; Campath-1H; Cytoxan; Etoposide; Fludarabine; Melphalan; Rituximab; Allogeneic Stem Cell Transplant; T-Cell Cell Adback; Natural Killer (NK) Cell Adback
MeSH Terms: conditions — Lymphoma; Leukemia; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma | interventions — Cytarabine; Carmustine; Alemtuzumab; Cyclophosphamide; Etoposide; fludarabine; fludarabine phosphate; Melphalan; Rituximab; Whole-Body Irradiation; Methotrexate; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NK Cell/T-Cell Infusion (Experimental): Possible Cell Adback - infusion NK cells or T-cells from donor given after blood stem cell transplantation for either Reduced intensity chemotherapy of campath, modified BEAM regimen of Campath-IH 15 mg intravenous (IV) Daily for 3 Days + BEAM Daily for 4 days (BCNU 300 mg/m^2 IV, Etoposide 100 mg/m^2 IV, Ara-C 100 mg/m^2 IV Daily for 4 days and Melphalan 100 mg/m^2 IV Over 30 Minutes for 1 Day) + Rituximab 375 mg/m^2 IV Over 5-7 Hours for 1 Day, followed by 1000 mg/m^2 IV Over 5-7 Hours Weekly for 3 Weeks]; or Non-myeloablative Preparative Regimen [Fludarabine 30 mg/m^2 IV Daily Over 1 Hour for 3 Days; Cyclophosphamide 1000 mg/m^2 IV Daily Over 1 Hour for 3 Days; Rituximab 375 mg/m^2 IV Over 5-7 Hours for 1 Day, followed by 1000 mg/m^2 IV Over 5-7 Hours Weekly for 3 Weeks; Campath-IH 15 mg IV Daily Over 30 Minutes for 3 Days; plus Total Body radiation (TBI)].
  Interventions: Drug: ARA-C; Drug: BCNU; Drug: Campath-1H; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Fludarabine; Drug: Melphalan; Drug: Rituximab; Other: Allogeneic Stem Cell Transplantation; Radiation: Total body radiation (TBI); Drug: Methotrexate; Drug: Tacrolimus; Procedure: Adback NK or T Cell

INTERVENTIONS:
Drug: ARA-C — 100 mg/m^2 IV Daily Over 1 Hour for 4 Days
  Other Names: Cytarbine; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: BCNU — 300 mg/m^2 IV Over 1 Hour for 1 Day
  Other Names: Carmustine; BiCNU
Drug: Campath-1H — 15 mg IV Daily Over 30 Minutes for 3 Days
  Other Names: Alemtuzumab; Campath
Drug: Cyclophosphamide — 1000 mg/m^2 IV Daily Over 1 Hour for 3 Days
  Other Names: Cytoxan; Neosar
Drug: Etoposide — 100 mg/m^2 IV Daily Over 3 Hours for 4 Days
  Other Names: VePesid
Drug: Fludarabine — 30 mg/m^2 IV Daily Over 1 Hour for 3 Days
  Other Names: Fludarabine Phosphate; Fludara
Drug: Melphalan — 100 mg/m^2 IV Over 30 Minutes for 1 Day.
Drug: Rituximab — 375 mg/m^2 IV Over 5-7 Hours for 1 Day, followed by 1000 mg/m^2 IV Over 5-7 Hours Weekly for 3 Weeks.
  Other Names: Rituxan
Other: Allogeneic Stem Cell Transplantation — Stem Cell Infusion on Day 0.
Radiation: Total body radiation (TBI) — TBI on Day 5 following chemotherapy, before stem cell infusion.
Drug: Methotrexate — 5 mg/m2 IV on Days +1, +3, and +6.
Drug: Tacrolimus — 0.03 mg/kg/day IV starting on Day -2, to be given through day 60, tapered by 20% every week, then discontinue by day 90.
  Other Names: Prograf
Procedure: Adback NK or T Cell — Adback natural killer (NK) cells or T cells after transplantation to enhance full engraftment of donor cells. Cell adback after transplantation applies only if there is no active GVHD, and no previous episode of grade II-IV GVHD.

SUMMARY:
Primary objective:

* To determine the safety of adback T- or Natural Killer (NK) cells in patients with lymphoid malignancies receiving allogeneic stem cell transplantation with Campath-IH containing conditioning regimen.

Secondary objective:

* To determine the efficacy (disease-free-survival) of this strategy.

DETAILED DESCRIPTION:
NK Cells, T-Cells, and the Study Drugs:

NK and T-cells from a donor may decrease the risk of relapse (reappearance of disease) after stem cell transplantation. NK cells and T-cells are kinds of white blood cells. Both types of cells have the ability to fight infection and "kill" tumor cells in the body. NK cells are called "natural killers" because, unlike T-cells, NK cells do not need to be activated ("turned on") by an antigen (a foreign substance) in order to "attack" and "kill" tumor cells.

Screening Tests:

Before starting treatment on this study, "screening tests" will be performed to help the doctor determine eligibility to take part in this study.

* Physical exam.
* Blood drawn (about 6 1/2 to 8 tablespoons) for routine tests, to check the effects of the transplantation, and for a liver function test. This routine blood draw will also include a pregnancy test for women who are able to have children. To be eligible to take part in this study, the pregnancy test must be negative.
* Urine collected for routine tests.
* Bone marrow biopsy performed to check the status of the disease. To collect a bone marrow biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.
* Chest x-ray, computed tomography (CT) scans, and an electrocardiogram (ECG -- a test that measures the electrical activity of the heart).

Study Treatment:

Treatment will begin within 30 days after the screening visit. All of the study drugs will be given through a central venous catheter (CVC) that will be left in place throughout treatment. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure in more detail, and a signed separate consent form for this procedure is required

Before starting the chemotherapy in this study, 21 or more days must have elapsed since the last biological therapy, chemotherapy, radiotherapy, or other investigational therapy.

PATIENTS RECEIVING BEAM, CAMPATH-IH, AND RITUXIMAB AS CONDITIONING:

BEAM is designed to kill leukemia and lymphoma cells by inserting itself into the cell DNA (genetic material of cells).

Alemtuzumab is designed to attach to a foreign substance (antigen) that is found on certain immune cells, which may cause the cells to die.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

On Day 1, BCNU will be given over 1 hour.

On Days 2-5, Ara-C will be given over 1 hour and etoposide over 3 hours. This will be repeated every 12 hours during these 4 days.

On Days 2-4, alemtuzumab will be given over 30 minutes. Hydrocortisone and tacrolimus will be given by vein during this time to help prevent or ease side effects, such as chills, skin rash, and/or hives.

On Day 6, melphalan will be given over 30 minutes.

Rituximab will also be given over 5-7 hours, 13 days before the transplantation and then once a week for a total of 4 doses.

On Day 7, after completion of chemotherapy, the blood or marrow stem cells that were collected earlier will be transplanted (given to your body) through the CVC over 30-45 minutes. This is the standard treatment.

On Days +1, +3, and +6 after the stem cell infusion, methotrexate will be given by vein to help decrease the risk of graft-versus-host disease.

G-CSF (filgrastim) will be injected just under your skin once a day until the neutrophil (a type of white blood cell) counts recover.

About 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

FOR PATIENTS RECEIVING FLUDARABINE, CYCLOPHOSPHAMIDE, CAMPATH-IH, RITUXIMAB,AND TBI:

TBI is designed to damage the DNA (the genetic material of cells) of cancer cells, which may kill the cancer cells.

Alemtuzumab is designed to attach to a foreign substance (antigen) that is found on certain immune cells, which may cause the cells to die.

Cyclophosphamide is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Fludarabine is designed to make cancer cells less able to repair damaged DNA (the genetic material of cells). This may increase the likelihood of the cells dying.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

On Days 1-3, alemtuzumab will be given over 30 minutes, fludarabine over 1 hour, and cyclophosphamide over 1 hour. Hydrocortisone and tacrolimus will be given by vein during this time to help prevent or ease side effects, such as chills, skin rash, and/or hives.

Rituximab will also be given over 5-7 hours, 13 days before the transplantation and then once a week for a total of 4 doses.

On Day 5, after completion of chemotherapy, TBI will be given, and later on the same day, the blood stem cells that were collected earlier will be transplanted (given back to your body) through the CVC over 30-45 minutes. This is the standard treatment.

On Days +1, +3, and +6 after the stem cell infusion, methotrexate will be given by vein to help decrease the risk of graft-versus-host disease.

G-CSF (filgrastim) will be injected just under your skin once a day until the neutrophil (a type of white blood cell) counts recover.

About 80 patients will take part in this study. All will be enrolled at M. D. Anderson.

ALL PATIENTS:

Infusion of NK Cells and T-Cells:

A "boost" of NK cells or T-cells from a donor may be given after blood stem cell transplantation, depending on the disease status and the amount of donor cells in the blood.

If a complete remission (disappearance of cancer symptoms) is achieved at 3 months after transplantation with more than 80% donor T-cells, no additional T-cells will be given.

If donor T-cells are less than 80% in the blood, then a boost of NK cells or T-cells will be given. The type of cells given will depend on results of DNA testing that was done during the screening visit to check the presence of molecules that may be able to activate ("turn on") NK cells in a specific area of your DNA. The same type of cell infusion may be repeated 8 weeks later, if the percentage of donor T-cells does not reach 100% in the blood.

If active disease persists at 3 months after transplantation, 1 dose of rituximab will be given once a week, or NK cells or T-cells will be given between the second and third dose of rituximab. Infusion of NK cells or T-cells may be repeated every 6 weeks (up to 12 weeks), if the disease does not achieve complete remission with the first infusion of cells.

It will be required to stay in the hospital from about 2 weeks before the transplantation until about 2-3 weeks after the transplantation. The additional cells will be infused on an outpatient basis.

Epinephrine and antihistamines will be available at the bedside during the NK cell infusion to help treat any allergic reactions.

Study Visits:

It will be required to stay in the Houston area for about 100 days after the transplantation. During initial study visits, the following tests/procedures will be performed after the transplantation.

* Blood transfusions of blood and platelets as needed.
* Blood drawn (about 6 teaspoons) for routine tests.
* Blood drawn (about 6-10 tablespoons) to check the effects of the transplantation.
* Urine collected for routine tests.
* Imaging scans, such as the ones performed during the screening visit.
* Bone marrow biopsy performed, when it is necessary.

Between Days 25-35 after transplantation, and then at 3 months, CT scans, positron emission tomography (PET), routine blood draws (about 6 teaspoons), and a bone marrow biopsy/aspirate will be performed. These tests will be done to check the status of the disease.

Length of Study:

Length of time on this study up to about 3 years, unless the disease gets worse or any intolerable side effects are experienced.

Follow-up:

After Day 35, if the disease is in remission with 100% donor cells, an evaluation will be performed every 3 months during the first year and then every 6 months up to 3 years.

If the disease is not in remission by Days 90-100, CT scans, PET scans, routine blood tests (about 6 teaspoons), and a bone marrow biopsy/aspirate will be performed every 6-8 weeks (after each NK or T-cell infusion until remission is achieved ). Then, these tests will be repeated every 6 months.

This is an investigational study. All of the drugs used in this study are FDA approved and commercially available. The use of NK cells is not FDA approved and commercially available. The use of the drugs and NK cells together in this study is investigational.

ELIGIBILITY:
Inclusion Criteria:

1. Up to 70 years of age.
2. B-cell lymphoid malignancies (those with CD20 negative disease at their diagnosis will not receive rituximab): This includes CLL/small lymphocytic lymphoma, follicular lymphoma, mantle cell, diffuse large cell, Splenic lymphoma, Mucosa-Associated Lymphoid Tissue (MALT), lymphoplasmacytic lymphoma and Burkitt's lymphoma.
3. Patients in relapse or considered at high risk for relapse.
4. In order to increase the chance of KIR-mismatching between recipient and donor, a 9/10 matched (mismatched locus C ) unrelated donor would be preferable. If a mismatched donor is not available, then a fully-matched unrelated donor or other 9/10 matched unrelated donor will be considered.
5. A sibling donor who is 9/10 matched may also be allowed.
6. Zubrod PS </= 2.
7. Left ventricular ejection fraction (LVEF)>/= 40% with no uncontrolled arrythmias or symptomatic heart disease.
8. Forced expiratory volume in one second (FEV1), Forced Expiratory Volume (FVC) and Carbon Monoxide Diffusing Capacity (DLCO) >/= 50%.
9. Serum creatinine < 1.8 mg/dL. Serum bilirubin < 3 * upper limit of normal,
10. Aspartate aminotransferase (AST) < 3 * upper limit of normal.
11. Signed, written Internal Review Board (IRB)-approved informed consent.
12. Men and women of reproductive potential must agree to follow accepted birth control methods for the duration of the study. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

1. Past history of anaphylaxis following exposure to CAMPATH-IH or Rituximab
2. Patient with active Central Nervous System (CNS) disease.
3. Positive Beta human chorionic gonadotrophin (hCG) text in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization, or currently breast-feeding.
4. Known infection with HIV, HTLV-I, Hepatitis B, or Hepatitis C.
5. Patients with other malignancies diagnosed within 2 years prior to Study registration (except skin squamous cell carcinoma).
6. Active uncontrolled bacterial, viral or fungal infections.
7. Major surgical procedure or significant traumatic injury within 4 weeks prior to Study registration.
8. Serious, non-healing wound, ulcer, or bone fracture.
9. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Study registration.
10. History of Stroke within 6 months.
11. Myocardial infarction within the past 6 months prior to Study registration.
12. Uncontrolled chronic diarrhea.
13. A prior allogeneic transplant from the same donor. Is there an age limit? Yes

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 26, 2007 to April 24, 2009. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 22 patients enrolled in the study, none were eligible to receive the adback T-Cell or Natural Killer (NK) cells.
Period: Overall Study
Arm/Group | NK Cell/T-Cell Infusion
Started | 22
Completed | 0
Not Completed | 22
Not completed — Not eligible for Adback Infusion | 22

BASELINE CHARACTERISTICS:
Arm/Group | NK Cell/T-Cell Infusion
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: years] | 54 [34 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: 6-month Treatment Related Mortality (TRM)
Description: Number of participant deaths in 6 months of T- cell or Natural killer (NK) cell adback treatment.
Time Frame: 6 Months
Population: Of the 22 patients enrolled, none received the adback T-Cell or NK cells treatment.
Arm/Group | NK Cell/T-Cell Infusion
Number analyzed (Participants) | 0

2. Secondary Outcome: One-year Disease-free Survival (DFS)
Description: Efficacy (disease-free-survival) defined as number of participants still living, without disease progression following T- cell or Natural killer (NK) cell adback. One-year disease-free survival (DFS) time estimated using the Kaplan-Meier estimator. Patients who experience disease recurrence considered to be a treatment failure event.
Time Frame: 1 Year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Most frequent and most serious adverse events collected during participants' standard of care (1 year and 10 months), not investigational treatment related adverse events.
Description: Adverse events were not collected under the study design treatment as no participants received the Adback Infusion (treatment).
Arm/Group | NK Cell/T-Cell Infusion
Serious Adverse Events (participants affected / at risk) | 14/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NK Cell/T-Cell Infusion (N=22)
Neutrophils (ANC/AGC) (Blood and lymphatic system disorders) | 1 — Absolute neutrophil count (ANC)/Absolute granulocyte count (AGC)
Acute respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Fever, Neutropenic (Blood and lymphatic system disorders) | 2
Hypomagnesemia (Blood and lymphatic system disorders) | 2
Stomatitis (Skin and subcutaneous tissue disorders) | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 1
Mood Alteration (General disorders) | 1
Pain, Chest Wall (Investigations) | 1
Graft versus host disease (GVHD), Chronic (Infections and infestations) | 1
Infection, Neutropenic (other) (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No